CLINICAL TRIAL: NCT00735137
Title: Randomized Study of Pessary vs Standard Management in Women With Increased Chance of Premature Birth
Brief Title: Randomized Study of Pessary Versus Standard Management in Women With Increased Chance of Premature Birth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 07/HW/10; ISRCTN01096902
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Preterm Birth
Keywords: Twins; Short cervix; Preterm birth; Vaginal pessary
MeSH Terms: conditions — Premature Birth | interventions — Pessaries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (No Intervention): Expectant management in twin pregnancy
- B (Experimental): Vaginal pessary treatment in twin pregnancy
  Interventions: Device: Vaginal pessary (CE0482, MED/CERT ISO 9003 / EN 46003)
- C (No Intervention): Expectant management in singleton pregnancy with short cervix; Women with cervix <15 mm will be commenced on vaginal progesterone
- D (Experimental): Vaginal pessary treatment in singleton pregnancy with short cervix; Women with cervix <15 mm will be commenced on vaginal progesterone
  Interventions: Device: Vaginal pessary (CE0482, MED/CERT ISO 9003 / EN 46003)

INTERVENTIONS:
Device: Vaginal pessary (CE0482, MED/CERT ISO 9003 / EN 46003) — Inserted from randomization till 36-37 weeks of gestation
  Other Names: Vaginal pessary, CE0482, MED/CERT ISO 9003 / EN 46003
  Arms: B; D

SUMMARY:
The aim of the study is to determine the effect of cerclage pessary on the incidence of spontaneous delivery between randomization (at 20-24+6 weeks) and 33+6 weeks in asymptomatic women with singleton pregnancies found at routine mid-trimester screening to have a cervix of <25 mm in length and in twin pregnancies.

DETAILED DESCRIPTION:
Prematurity is responsible for more than half of all neonatal deaths and whilst advances in neonatal care have dramatically improved survival of extremely premature infants, there remains a significant risk of handicap and disability in survivors and an associated social and economic burden.

In singleton pregnancies the rate of spontaneous premature birth before 34 weeks is about 1% and the risk of spontaneous early delivery is inversely related to cervical length. The group with cervix of 1-15 mm accounted for 28% of all spontaneous deliveries before 34 weeks and those with cervix of 16-25 mm accounted for 21%. The rate of spontaneous premature birth before 34 weeks is about 13% in twin pregnancies.

Potential methods for the prevention of preterm delivery include bed rest, cervical cerclage and prophylactic administration of progesterone. The prophylactic administration of progesterone beginning in mid-gestation to women who previously had a premature birth and in those with a short cervix has been shown to reduce the rate of spontaneous preterm birth before 34 weeks. On the other hand, randomized studies reported that, in twin pregnancies, bed rest was associated with a significant increase, rather than decrease, in the rate of early preterm delivery.

There is some evidence that the rate of premature birth can be dramatically reduced by the insertion of a vaginal pessary (cerclage pessary, CE0482, MED/CERT ISO 9003 / EN 46003).

This will be a multicenter trial in the UK and other countries. During routine ultrasound scan at 20-24 weeks of gestation for examination of fetal anatomy and growth, all women with twin pregnancy or with singleton pregnancy found to have a cervix of <25 mm in length and where the fetuses are found to be alive with no major abnormalities, severe twin to twin transfusion syndrome or severe fetal growth restriction in one of the fetuses (in the case of twin pregnancy), will be invited to participate in a randomized trial of standard management vs vaginal insertion of a cerclage pessary. For singleton pregnancy, in both arms the patients with cervical length <15 mm will be given prophylactic progesterone (200 mg vaginal capsule per night up to 34 weeks). Randomization and insertion of the pessary (in those allocated to this group) will be carried out within 5 days after the 20-24 weeks scan.

The pessary will be removed by a simple vaginal examination at 37 weeks or earlier before medically indicated preterm induction of labor or elective cesarean section. The pessary will also be removed in women in preterm labor not responding to tocolytic therapy. In monochorionic twins some obstetricians advise that delivery is carried out at around 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Women with singleton pregnancies and with a cervical length of 25 mm or less
2. Women with twin pregnancies

Exclusion Criteria:

1. Major fetal abnormalities (defined as those that are lethal or require prenatal or postnatal surgery), fetal death, severe twin to twin transfusion syndrome or severe fetal growth restriction in one of the fetuses (in the case of twin pregnancy) diagnosed before randomization.
2. Painful regular uterine contractions, history of ruptured membranes, or prophylactic cerclage before randomization.
3. Patients who are unconscious, severely ill, mentally handicapped or under the age of 16 years.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2109 (Actual)
Dates: Start 2008-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be spontaneous delivery from randomization to 33 weeks and 6 days (237 days) of gestation. | 10 weeks

SECONDARY OUTCOMES:
Low birth weight; Fetal or neonatal death; Major adverse outcomes (IVH, RDS, retinopathy of prematurity or necrotizing enterocolitis); Need for neonatal special care (ventilation, phototherapy, treatment for sepsis, blood transfusion) | Within the first year

CONTACTS AND LOCATIONS:
Overall Officials: Kypros H Nicolaides, Professor, Study Director — Consultant,Director of the Department of Fetal Medicine
Locations (24):
- Medical University of Vienna-department of Obstetrics and Gynaecology, Vienna, Austria
- Brazil (2):
  - Universidade Federal Fluminense - Hospital Universitário Antônio Pedro, Niterói, Rio de Janeiro
  - University of Campinas, São Paulo
- Hospital Clinico Universidad de Chile, Santiago, Chile
- Colombia (2):
  - Hospital San Jose, Bogotá
  - Hospital Universitario San Vicente de Paúl, Medellín
- Virchow Clinic Charite, Berlin, Germany
- Chinese University of Hong Kong, Hong Kong, Hong Kong
- Fernandez Hospital, Bogulkunta,, Bogulkunta, India
- Ospedale Valduce, Como, Lombardy, Italy
- Portugal (2):
  - Maternidade Dr. Alfredo da Costa, Lisbon
  - Hospital San Teotonio, Viseu
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- Spain (3):
  - Hospital Universitario Materno Infantil de Canarias, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Universitario Virgen de las Nieves, Granada
  - Virgen de La Arrixaca, Murcia
- United Kingdom (8):
  - Heatherwood and Wexham Park Hospitals, Wexham Park Hospital, Slough, Berkshire
  - Barking, Havering and Redbridge Hospitals NHS Trust, Romford, Essex
  - Southend Hospital NHS Trust, Essex
  - The Medway Maritime Hospital NHS Trust, Kent
  - University College London Hospitals NHS Foundation Trust, London
  - The Lewisham Hospital NHS Trust, London
  - Queen Elizabeth Hospital NHS Trust, London
  - King's College Hospital NHS Trust, London